CLINICAL TRIAL: NCT06287788
Title: The Prediction of a Mucosal Contouring Method Based on Swallowing-induced Breakthrough Pain for Radiation-induced Oropharyngeal Mucositis in Patients With Nasopharyngeal Carcinoma: an Observational Study
Brief Title: A Mucosal Contouring Method Based on Swallowing-induced Breakthrough Pain for Radiation-induced Oropharyngeal Mucositis
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-068
Record Dates: First submitted 2024-02-17; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Radiation-induced Oropharyngeal Mucositis; Swallowing-induced Breakthrough Pain
Keywords: Nasopharyngeal carcinoma; Radiation; Oropharyngeal mucositis; Swallowing-induced breakthrough pain; Delineation method
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The performance of the predictive models for severe oropharyngeal mucositis established using current oral mucosal contouring method was unsatisfactory in nasopharyngeal carcinoma (NPC). Whereas the predictive model of a mucosal contouring method based on swallowing-induced breakthrough pain exhibited better overall performance. The aim of this prospective, multicenter, observational study was to further explore the predictive efficacy of this mucosal delineation method for radiation-induced oropharyngeal mucositis in NPC.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is particularly prevalent in southern China. Radiation-induced oropharyngeal mucositis is one of the most common acute toxicities in patients with NPC receiving radiotherapy. Swallowing-induced breakthrough pain is a prominent clinical challenge for radiation-induced oropharyngeal mucositis, which has a great impact on patients' quality of life and treatment outcomes. Nonetheless, no particularly effective therapeutic methods or medication are available currently, thus making timely and accurate prediction, identifying high-risk patients, and providing appropriate interventions are critical in reducing or delaying the occurrence of severe oropharyngeal mucositis. It has been found that the performance of the predictive models for severe oropharyngeal mucositis established using either oral cavity contouring method or mucosa surface contouring method was unsatisfactory in NPC. The investigators defined a delineation method based on the mucosal areas of radiation-induced injury resulting in swallowing-induced breakthrough pain in locally advanced NPC, and our preliminary results demonstrated that the predictive model exhibited better overall performance. Therefore, the investigators aimed to conduct a prospective, multicenter, observational study to further explore the predictive efficacy of this mucosal delineation method for radiation-induced oropharyngeal mucositis in NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed written consent.
2. Age ≥ 18 years.
3. Histologically confirmed as nasopharyngeal carcinoma, and currently undergoing radical radiotherapy or chemoradiotherapy.
4. Complete and continuous records of oral / oropharyngeal mucositis grading, and self-reported swallowing-induced breakthrough pain.

Exclusion Criteria:

1. Existence of poor oral hygiene, untreated dental or periodontal diseases, and metal dental restorations.
2. Current untreated or unresolved conditions like unstable heart diseases requiring treatment, and poorly controlled diabetes mellitus.
3. Body mass index (BMI) <18.5.
4. Unsuitable to participate in current study, according to researchers' assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nasopharyngeal carcinoma after receiving radical radiotherapy or chemoradiotherapy
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The AUC of the predictive model | Through study completion, up to 3 years
  The area under the ROC (receiver operating characteristic) curve (AUC) of the predictive model

SECONDARY OUTCOMES:
The accuracy, sensitivity, specificity, positive predictive value, negative predictive value and F1 score of the predictive model | Through study completion, up to 3 years
  To obtained these metrics, true positive (TP), false positive (FP), true negative (TN), and false negative (FN) were calculated from the confusion matrix.
  Sensitivity = TP/(TP + FN) Specificity = TN/(TN + FP) Accuracy = (TP+TN)/(Σ Total population) Positive Predictive value (PPV) = TP/(TP + FP) Negative Predictive value (NPV) = TN/(TN + FN) F1 score = 2TP/(2TP + FP + FN)
The important predictors of severe oropharyngeal mucositis in the predictive model | Through study completion, up to 3 years
  The importance of variables included in the predictive model was measure, and those with a higher value indicating a greater contribution to the model's classification accuracy were viewed as the important predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Guan, Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No